CLINICAL TRIAL: NCT04123704
Title: A Phase II Study of Sitravatinib in Metastatic, Pre-treated, Triple Negative Breast Cancer
Brief Title: Sitravatinib in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor due to lack of interest
Sponsor: Xiang Zhang (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Xiang Zhang, Professor, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43432
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Stage IV; Triple Negative Breast Cancer; Breast Neoplasms; Breast Cancer Metastatic
Keywords: triple negative; metastatic breast cancer; sitravatinib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sitravatinib (Experimental): Sitravatinib 100 mg daily
  Interventions: Drug: Sitravatinib

INTERVENTIONS:
Drug: Sitravatinib — sitravatinib capsule
  Other Names: MGCD516

SUMMARY:
This study evaluates the efficacy of sitravatinib in patients with metastatic breast cancer. All study participants will receive sitravatinib, 100 mg daily, until their cancer worsens, or until they develop intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Women or men age 18 and older
* Metastatic or locally advanced inoperable breast cancer (beyond curative management) that is measurable according to RECIST 1.1 criteria. Note: Patients with bone-only disease are eligible if there is at least 1 lytic lesion that can be followed for response.
* Tumor is estrogen receptor (ER) negative and progesterone receptor (PR) negative per the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) Guidelines of 2010.
* Tumor is HER2neu negative per ASCO/CAP Guidelines of 2018
* Patient has archival tissue from metastatic or locally advanced breast cancer for the analysis of PTPN12 status
* At least one prior line of chemotherapy with or without a PD-L1 or PD-1 antibody in the metastatic setting
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count > 1000/mcL
  * Hemoglobin > 11 g/dL
  * Platelets > 100,000/mcL
  * Total bilirubin < 1.5 X normal institutional limits
  * Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 2.5 X institutional ULN or ≤ 5.0 × ULN for patients with documented liver metastases.
  * Creatinine within normal institutional limits
  * Creatinine clearance ≥ 30 mL/min
  * Normal left ventricular ejection (LVEF) function defined as normal left ventricular wall motion and ejection fraction of ≥ 50%.
* If patient has brain metastasis, documented treatment and stability for at least 30 days by scans and off steroids at the time of enrollment
* Women of child bearing age and actively menstruating must have a negative pregnancy test prior to starting study treatment.
* If sexually active in a way that could lead to pregnancy, participant must agree to use a highly effective method of birth control starting at the time of informed consent and continuing throughout the study and for at least 3 months after the final dose of sitravatinib.
* Ability to understand and the willingness to give informed consent

Exclusion Criteria:

* Uncontrolled hypertension defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100, on two or more occasions within 30 days prior to enrollment.
* Imaging suggestive of Lymphangitic carcinomatosis in the lung, or use of home oxygen
* Untreated brain metastases.
* Women who are pregnant or nursing
* Concurrent metastatic disease of another tumor type
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of sitravatinib
* History of stroke, pulmonary embolus (PE), or myocardial infarction (MI)
* Known proteinuria of ≥ 2 g urinary protein/24 h
* HIV-positive participants
* History of Hepatitis C or Hepatitis B infection
* History of congestive heart failure (CHF), and/or LVEF less than 50%
* Concurrent use of medications that prolong QTc (listed in Section 9, Table 11). These medications need to be discontinued at least 2 weeks prior to starting study treatment.
* Concurrent medical condition that, in the sole judgment of the principal investigator, would make the patient inappropriate for trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Kent Osborne, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sitravatinib
Started | 3
Completed | 1 (1 patient reached the primary outcome milestone of progression-free survival at 24 weeks.)
Not Completed | 2
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Progression-Free Survival at 24 Weeks (PFS24)
Description: Progression-free survival 24 weeks after starting study treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Progressive Disease, >=20% increase in the sum of the smallest diameter of target lesions, or appearance of one or more new lesions.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
percentage of participants | 33.3 [0.8 to 90.6]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the duration of time from initiation of study treatment until progression. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Progressive Disease, >=20% increase in the sum of the smallest diameter of target lesions, or appearance of one or more new lesions.
Time Frame: Up to 16 months
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
weeks | 24.6 (16.3)

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants who achieve a Complete Response (CR) or Partial Response (PR) to treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 16 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
percentage of participants | 33.3 [0.8 to 90.6]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate is defined as the percentage of participants who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither >=30% decrease in sum of longest diameter of target lesions nor >=20% increase in sum of shortest diameter of target lesions.
Time Frame: Up to 16 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
percentage of participants | 66.7 [9.4 to 99.2]

5. Secondary Outcome: Number of Participants With Grade 3 or Higher AEs
Description: Adverse events will be assessed and graded per the NCI CTCAEv5.
Time Frame: Up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were assessed starting at beginning of treatment until 30 days after disease progression or at study completion (up to 16 months), whichever comes first. All-cause mortality was assessed at study completion (up to 16 months from the treatment start date).
Arm/Group | Sitravatinib
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib (N=3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib (N=3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT04123704/Prot_SAP_000.pdf